CLINICAL TRIAL: NCT00831779
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Trial to Evaluate the Effects of Dapagliflozin on Insulin Resistance and Insulin Secretion in Subjects With Type 2 Diabetes
Brief Title: Effects of Dapagliflozin on Insulin Resistance and Insulin Secretion in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Astra Zeneca, Bristol-Myers Squibb (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB102-045
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental)
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 5 mg, once daily, 12 weeks
  Other Names: BMS-512148
  Arms: Dapagliflozin
Drug: Placebo — Tablets, Oral, 0 mg, Once daily, 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of dapagliflozin on insulin sensitivity

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes and inadequate glycemic control, defined as A1C ≥ 7.0 and ≤ 10.0% at the enrollment visit
* Subjects should have been receiving either metformin therapy OR metformin therapy AND one insulin secretagogue for at least 12 weeks prior to enrollment
* C-peptide ≥ 1.0 ng/ml (0.34 nmol/l)
* BMI ≤ 45.0 kg/m2

Exclusion Criteria:

* Urine albumin to creatinine ratio (UACR) > 1,800 mg/g (203.4 mg/mmol/Cr)
* Aspartate Aminotransferase (AST) > 3X Upper limit of normal (ULN)
* Alanine aminotransferase (ALT) > 3X ULN
* Serum Total Bilirubin > 2 mg/dL (34.2 μmol/l)
* Serum Creatinine (Scr) ≥ 1.50 mg/dL (133 μmol/l) for men; SCr ≥ 1.40 mg/dL (124 μmol/l) for women
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncological, endocrine, psychiatric, or rheumatic diseases

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Va San Diego Healthcare System, San Diego, California
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Temple University General Clinical Research Center, Philadelphia, Pennsylvania

REFERENCES:
- See also: Publication — http://online.liebertpub.com/doi/full/10.1089/dia.2013.0167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 116 participants enrolled, 50 completed a qualification period. Of these 50 participants, 44 were randomized and received treatment. Of these 44 participants, 42 completed double-blind treatment period.
Groups:
- Placebo + Background Anti-Diabetes Medication: Placebo tablets, oral, once daily, 12 weeks
- Dapagliflozin 5 mg + Background Anti-Diabetes Medication: Dapagliflozin tablets, oral, once daily, 12 weeks
Period: Overall Study
Arm/Group | Placebo + Background Anti-Diabetes Medication | Dapagliflozin 5 mg + Background Anti-Diabetes Medication
Started | 21 | 23
Completed | 20 | 22
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — No longer met criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Background Anti-Diabetes Medication | Dapagliflozin 5 mg + Background Anti-Diabetes Medication | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.3 (8.02) | 56.2 (8.85) | 54.8 (8.49)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 18 | 19 | 37
  65-70 years | 3 | 4 | 7
Sex/Gender, Customized [Number; unit: Participants]
  Male | 14 | 15 | 29
  Female | 7 | 8 | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 15 | 13 | 28
  Black/African American | 6 | 9 | 15
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Percent Change From Baseline in Insulin Sensitivity at Week 12 (Last Observation Carried Forward [LOCF])
Description: Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Measurements were obtained during the randomization visit and Week 12 in the double-blind period.
Time Frame: From Baseline to Week 12
Population: All randomized participants who received study medication and had nonmissing values at baseline and Week 12 (LOCF)
Measure: Mean (Standard Error); unit: % Change of Baseline Insulin Sensitivity
Arm/Group | Placebo + Background Anti-Diabetes Medication | Dapagliflozin 5 mg + Background Anti-Diabetes Medication
Number analyzed (Participants) | 19 | 22
% Change of Baseline Insulin Sensitivity | -9.99 (4.0392) | 7.98 (4.4849)
Statistical Analysis 1: Comparison: Placebo + Background Anti-Diabetes Medication vs Dapagliflozin 5 mg + Background Anti-Diabetes Medication; Test type: Superiority or Other; p = 0.0059, ANOVA — Primary endpoint was tested at alpha=0.05; Mean Difference (Final Values) = 19.97, 95% CI 2-sided [5.75 to 36.10], Standard Error of Mean 7.4685

2. Secondary Outcome: Adjusted Mean Change From Baseline in Insulin Secretion at Week 12 (Last Observation Carried Forward [LOCF])
Description: as for outcome 1
Time Frame: From Baseline to Week 12
Population: All randomized participants who received study medication and had nonmissing values at baseline and Week 12 (LOCF)
Measure: Mean (Standard Error); unit: mU/L*min
Arm/Group | Placebo + Background Anti-Diabetes Medication | Dapagliflozin 5 mg + Background Anti-Diabetes Medication
Number analyzed (Participants) | 19 | 23
mU/L*min | -12.73 (10.7107) | 15.39 (9.5930)
Statistical Analysis 1: Comparison: Placebo + Background Anti-Diabetes Medication vs Dapagliflozin 5 mg + Background Anti-Diabetes Medication; Test type: Superiority or Other; p = 0.0598, ANOVA — Secondary endpoint was tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = 28.13, 95% CI 2-sided [-1.22 to 57.48], Standard Error of Mean 14.4984

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of double-blind treatment 12 weeks plus 4 days for non-serious adverse event; plus 30 days for serious adverse event.
Arm/Group | Placebo + Background Anti-Diabetes Medication | Dapagliflozin 5 mg + Background Anti-Diabetes Medication
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 8/21 | 9/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Background Anti-Diabetes Medication (N=21) | Dapagliflozin 5 mg + Background Anti-Diabetes Medication (N=23)
HEADACHE (Nervous system disorders) | 3 (4) | 3 (4)
INFUSION SITE PAIN (General disorders) | 1 (2) | 2 (2)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 2 (2)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 1 (2)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No